CLINICAL TRIAL: NCT02353481
Title: 1 Year Post Discharge Prognostic Model From the National Heart Failure Audit (NHFA)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: National Institute for Cardiovascular Outcomes Research (Other); British Society for Heart Failure (Unknown)
Responsible Party: Principal Investigator, Aminat J Shote, Information Analyst, University College London, University College, London
Other Study IDs: NICOR-Heart Failure
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure: All patients in the audit that meets the eligibility criteria
  Interventions: Other: Heart Failure Management

INTERVENTIONS:
Other: Heart Failure Management

SUMMARY:
The aim of the study is to develop and assess a prognostic model for patient's survival up to 1 year after unscheduled acute heart failure hospital admission in England and Wales.

DETAILED DESCRIPTION:
There is a need for a prognostic model for 1 year survival of patients discharged alive after an unscheduled hospital admission for heart failure. This study aims to develop and validate a prognostic model that will enable management planning and facilitate the identification of therapeutic needs or targets. Also, it will assist care providers to predict or quantify patients' survival based on their baseline characteristics.

The National Heart Failure Audit (NHFA) held by National Institute for Cardiovascular Outcomes Research (NICOR) is one of the largest available national heart failure registry. It includes data from unscheduled heart failure admissions in England and Wales. In the audit, heart failure diagnosis is defined as a diagnosis that has been confirmed by imaging or brain natriuretic peptide (BNP) measurement. This study will use NHFA data to develop and validate the proposed model.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and above
* survived to discharge
* have mortality status at 1 year post-discharge

Exclusion Criteria:

Non-index heart failure admissions during the study period will be excluded from the study sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unscheduled heart failure admissions in England and Wales are recorded in the National Heart Failure Audit. Therefore, patients with data in the audit will be eligible for inclusion if they meet the inclusion criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 63320 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

REFERENCES:
- [Background] Pocock SJ, Wang D, Pfeffer MA, Yusuf S, McMurray JJ, Swedberg KB, Ostergren J, Michelson EL, Pieper KS, Granger CB. Predictors of mortality and morbidity in patients with chronic heart failure. Eur Heart J. 2006 Jan;27(1):65-75. doi: 10.1093/eurheartj/ehi555. Epub 2005 Oct 11. PMID 16219658
- [Background] Adams KF Jr, Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP; ADHERE Scientific Advisory Committee and Investigators. Characteristics and outcomes of patients hospitalized for heart failure in the United States: rationale, design, and preliminary observations from the first 100,000 cases in the Acute Decompensated Heart Failure National Registry (ADHERE). Am Heart J. 2005 Feb;149(2):209-16. doi: 10.1016/j.ahj.2004.08.005. PMID 15846257
- [Background] Levy WC, Mozaffarian D, Linker DT, Sutradhar SC, Anker SD, Cropp AB, Anand I, Maggioni A, Burton P, Sullivan MD, Pitt B, Poole-Wilson PA, Mann DL, Packer M. The Seattle Heart Failure Model: prediction of survival in heart failure. Circulation. 2006 Mar 21;113(11):1424-33. doi: 10.1161/CIRCULATIONAHA.105.584102. Epub 2006 Mar 13. PMID 16534009
- [Background] Pocock SJ, Ariti CA, McMurray JJ, Maggioni A, Kober L, Squire IB, Swedberg K, Dobson J, Poppe KK, Whalley GA, Doughty RN; Meta-Analysis Global Group in Chronic Heart Failure. Predicting survival in heart failure: a risk score based on 39 372 patients from 30 studies. Eur Heart J. 2013 May;34(19):1404-13. doi: 10.1093/eurheartj/ehs337. Epub 2012 Oct 24. PMID 23095984